CLINICAL TRIAL: NCT05733845
Title: Evaluation of Molecular Mechanisms of Non-response to Treatments, Relapses and Remission in Ulcerative Colitis and Crohn's Disease Patients Receiving First Time Standard of Care Biological Treatment
Brief Title: Evaluation of Molecular Mechanisms of Non-response to Therapy in Patients With Inflammatory Bowel Disease
Acronym: 3TR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Dr Laurent PEYRIN-BIROULET, Doctor, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A02277-36
Record Dates: First submitted 2023-01-16; First posted 2023-02-17 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: biomarkers; Crohn's disease; ulcerative colitis; disease activity; therapy reponse
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — Sampling Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Samples (Other): The intervention is to collect blood; urine; saliva and stool samples but also mucosal biopsies at each protocol visits (baseline and follow up visits).
  Interventions: Other: Samples

INTERVENTIONS:
Other: Samples — The intervention is to collect blood; urine; saliva and stool samples but also mucosal biopsies at each protocol visits (baseline and follow up visits).

SUMMARY:
Inflammatory bowel diseases (IBD) represent a group of immune-mediated disorders, in which currently unidentified trigger factors drive the manifestation of chronic relapsing- remitting destructive inflammatory episodes in the gut. IBD comprise two main disease entities, ulcerati\ie colitis (UC) and Crohn s disease (CD). The diseases differ in anatomical distribution, with continuous, uniform inflammation restricted to the colon in UC, and multifocal inflammation extended throughout the entire gastrointestinal tract from mouth to anus in CD. Clinical symptoms of IBD may include bloody stools, abdominal pain, fatigue, diarrhoea, fever and weight loss. Extra-intestinal symptoms occurring in up to 40% of patients, e.g. anaemia, skin lesions (e.g. erythema nodosum, pyoderma), arthritis and uveitis, and other complications directly related to the disease organ, such as fistula in CD are considered to reflect an overwhelming systemic inflammatory state. Disease onset typically manifests at age 15-35 years, men and women are almost equally affected. In addition, paediatric forms of IBD that often represent complex, se\/ere monogenic forms of the disease, are seen. The incidence rates of IBD in Europe are about 6.3 (CD) and 11.8 (UC) per 100.000 persons. With growing incidence rates and overall reduced mortality the lifetime prevalence of IBD is expected to rise. The estimated lifetime prevalence of 0.3%-0.5% of the European population corresponds to estimates of 1.5-2 million patients with IBD.

Appropriate selection of therapies and their timing of introduction (decision support) in the course of IBD will be essential to reach a higher degree of disease control (across patients and within individual patients) than it is achie\led today. In many instances, comparati\ie data is missing and combinations or sequential therapies are not developed. In summary, despite some treatment successes, major challenges remain.

The investigators have decided to include patients with inflammatory bowel disease (IBD) in which targeted therapies are administered as part of standard helathcare and which aims at identifiyng solid biomarker signatures as well as molecular pathways and mechanisms linked to response and non-response to therapy. Choice od medications (which are all approved for first line use) is by treating physicians. All follow-up procedures are according to standards of care.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 18 years of age (at the time of signing the Informed Consent)
* Person informed about study organization and having signed the informed consent.
* Established diagnosis of Crohn's dsease or ulcerative colitis with a minimum disease duration of 3 months
* Moderate to severe disease activity

  * UC : Mayo Score ≥ 6 including endoscopy score of ≥ 2
  * CD : CDAI score betwenn 220 and 450 (inclusive)
* Indication to start any biological or small molecule agent (anti-TNF, anti-IL 21/23, anti-integrin and JAK-inhibitors)
* In case of treatment with corticosteroid : stable dose for at least 3 weeks prior to baseline, dosage ≤ 20 mg prednisone
* Indication for colonoscopy for the assessment of disease activity as for standards of care and current guidelines
* Person affiliated to or beneficiary of a social security plan

Exclusion Criteria:

* Diagnosis of indeterminate colitis, microscopic colitis, ischaemic colitis, infectious colitis, radiation colitis
* Absolute contraindications to colonoscopy procedures, complication during previous endoscopy
* Bleeding disorders
* Indication for surgery for UC
* Rectal topical therapy (enemas or suppositories) ≤ 2 weeks prior to baseline
* Treatment with > 20 mg prednisone within 3 weeks prior to baseline
* Anaemia (haemoglobbin < 10g/dl) at baseline
* Subject unable to comply with the study procedures
* Person referred in articles L.1121-5, L. 1121-7 and L.1121-8 of the Public Health Code:

  * Pregnant, parturient or breastfeeding woman
  * Minor person (non-emancipated)
  * Adult person under legal protection (any form of public guardianship)
  * Adult person incapable of giving consent and not under legal protection
* Person deprived of liberty for judicial or administrative decision, person under psychiatric care as referred in articles L. 3212-1 and L. 3213-1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2030-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
To identify solid biomarkers signatures as well as molecular pathways and mechanisms linked to response and non-response to therapy in ulcerative colitis patient. | week 14
  -For Ulcerative Colitis (UC) patient: overall Mayo score correlated with Mayo endoscopy and bleeding subscore will be measured.
  Mayo score composed by 4 items: stool frequency; rectal bleeding, mucosal appearance at endoscopy and physician rating of disease activity.
  Mayo score:
  Score <2 : no activity Score between 3 and 5: mild activity Score between 6 and 10 :moderate activity Score >11 : severe activity
To identify solid biomarkers signatures as well as molecular pathways and mechanisms linked to response and non-response to therapy in Crohn's disease patient. | week 14
  -For Crohn's Disease (CD) patient : Crohn's disease activity index (CDAI) and simple endoscopic response (SES-CD) wil be measured.
  CDAI is the sum of 8 components: number of liquid or soft stools, daily abdominal pain, patient well-being, complications, use of diphenoxylate or opiates as anti-diarreheal, abdominal mass, hematocrit and body weight.
  Level of disease activity:
  Non-active disease: CDAI < 150 Mild disease activity: CDAI >= 150 and <220 Moderate disease activity: CDAI >= 220 and <450 Severe disease activity: CDAI > 450
  SES-CD assesses the size of mucosal ulcers, the ulcerated surface, the endoscopic extension and the presence of stenosis.
  SES-CD score:
  0 - 2 remission 3 - 6 mild endoscopic activity 7 - 15 moderate endoscopic activity > 15 severe endoscopic activity

SECONDARY OUTCOMES:
To correlate identifed potential biomarkers with disease activity, progression and response to therapy by clinical remission in Crohn's disease patient | week 52
  Remission will be evaluated by mucosal healing (simple endoscopic response (SES-CD)).
  SES-CD assesses the size of mucosal ulcers, the ulcerated surface, the endoscopic extension and the presence of stenosis.
  SES-CD score:
  0 - 2 remission 3 - 6 mild endoscopic activity 7 - 15 moderate endoscopic activity > 15 severe endoscopic activity
To correlate identifed potential biomarkers with disease activity, progression and response to therapy by clinical remission in Ulcerative colitis patient | week 52
  Remission will be evaluated by mucosal healing (Mayo score). Mayo score composed by 4 items: stool frequency; rectal bleeding, mucosal appearance at endoscopy and physician rating of disease activity.
  Mayo score:
  Score <2 : no activity Score between 3 and 5: mild activity Score between 6 and 10 :moderate activity Score >11 : severe activity
To correlate identifed potential biomarkers with disease activity, progression and response to therapy by patient-reported outcomes | week 52
  Symptomatic remission assessed by patient-reported outcomes
To correlate identifed potential biomarkers with disease activity, progression and response to therapy by complications-reported. | week 52
  Complications-reported: hospitalizations due to inflammatory-bowel disease; treatment intensification including introduction of toxic long-term therapies (i.e. systemic glucocorticoids); presence of new stenosis; presence of new fistula ;new infections or intestinal surgery known
To correlate identifed potential biomarkers with disease activity, progression and response to therapy by disease progression. | week 52
  Presence of flares e.g.

OTHER OUTCOMES:
Fatigue assessment | Baseline visit (time -4 weeks to 0), visit 1 (time 0), visit 2 (time 0+2 weeks), visit 3 (time 0+14 weeks), visit 4 (time 0+26 weeks) and visit 5 (time 0+52 weeks)
  Evaluated by Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F).
  FACIT-F is a 40-items measure that assesses self-reported fatigue and its impact upon daily activites and function.
  5 point Likert-type scale. Subscale domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, Fatigue Minimum value: 0 = better outcome Maximum value: 160= worst outcome
Emotional distress-depression assessment | Baseline visit (time -4 weeks to 0), visit 1 (time 0), visit 2 (time 0+2 weeks), visit 3 (time 0+14 weeks), visit 4 (time 0+26 weeks) and visit 5 (time 0+52 weeks)
  Evaluated by Patient-Reported Outcomes Measurement Information System® (PROMIS®) Depression scale.
  PROMIS-Depression is a 8-items scale. Score between 8 and 40. 8= best health statein the past 7 days. 40= worst health state in the past 7 days.
General Health Survey assessment | Baseline visit (time -4 weeks to 0), visit 1 (time 0), visit 2 (time 0+2 weeks), visit 3 (time 0+14 weeks), visit 4 (time 0+26 weeks) and visit 5 (time 0+52 weeks)
  Evaluated by the The Short Form (36) Health Survey (SF36). SF36 is a patient-reported survey of patient health that covers physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions.
  Score range from 0 to 100. 100= more favorable health state. 0= worst health state.
Health status assessment | Baseline visit (time -4 weeks to 0), visit 1 (time 0), visit 2 (time 0+2 weeks), visit 3 (time 0+14 weeks), visit 4 (time 0+26 weeks) and visit 5 (time 0+52 weeks)
  Evaluated by the 5-level EQ-5D version (EQ-5D-5L). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
  Score between 5 and 25. 5=best health state 25= worst health state
  The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  100= best health state 0= worst health state.
Medical complications | Until week 104
  Long-term outcome (complications until week 104). Complication like stenosis, fistula, development of PSC, infections, flares, hospitalizations, treatment intensification including introduction of toxic long-term therapies (i.e. systemic glucocorticoids) or intestinal surgery will be documented during the entire observational period.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent PEYRIN-BIROULET, Principal Investigator — CHRU of Nancy, Hepatogastroenterology Department
Locations (1):
- CHRU of Nancy, Vandœuvre-lès-Nancy, CHRU de Nancy, France

REFERENCES:
- [Result] Burisch J, Jess T, Martinato M, Lakatos PL; ECCO -EpiCom. The burden of inflammatory bowel disease in Europe. J Crohns Colitis. 2013 May;7(4):322-37. doi: 10.1016/j.crohns.2013.01.010. Epub 2013 Feb 8. PMID 23395397
- [Result] Ng SC, Shi HY, Hamidi N, Underwood FE, Tang W, Benchimol EI, Panaccione R, Ghosh S, Wu JCY, Chan FKL, Sung JJY, Kaplan GG. Worldwide incidence and prevalence of inflammatory bowel disease in the 21st century: a systematic review of population-based studies. Lancet. 2017 Dec 23;390(10114):2769-2778. doi: 10.1016/S0140-6736(17)32448-0. Epub 2017 Oct 16. PMID 29050646